CLINICAL TRIAL: NCT04926155
Title: A Prospective, Randomized Trial Comparing Metformin Plus Androgen Deprivation Therapy (ADT) and Abiraterone With ADT Plus Abiraterone in Metastatic Castration-resistant Prostate Cancer
Brief Title: The Effect of Metformin in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonghong Li, Prinicipal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-072
Record Dates: First submitted 2021-06-11; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Prostate Cancer
Keywords: mCRPC; abiraterone; metformin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin+ADT+abiraterone (Experimental): Patients in this arm will be treatet with metformin plus ADT and abiraterone
  Interventions: Drug: Metformin
- ADT+abiraterone (No Intervention): Patients in this arm will be treatet with ADT and abiraterone, Abiraterone 1000mg once daily until disease progression.

INTERVENTIONS:
Drug: Metformin — The starting daily dose of metformin is 500mg once daily, and add a dose of 500mg per week until the target dose of 2000mg once daily if tolerated. Metformin will be continued until disease progression.
  Other Names: Metformin Hydrochloride Sustained Release Tablets
  Arms: Metformin+ADT+abiraterone

SUMMARY:
The purpose of this study is to assess the effect of the addition of metformin to abiraterone on survival in patients with metastatic castration-resistant prostate cancer (mCRPC). The half the patients will receive metformin in combination with androgen deprivation therapy (ADT) and abiraterone, and the other half will receive ADT and abiraterone only.

DETAILED DESCRIPTION:
Metastatic castration-resistant prostate cancer (mCRPC) can be treated with ADT plus abiraterone, ADT plus enzalutamide, ADT plus cabazitaxel, ADT plus docetaxel, ADT plus olaparib. However, patients have short overall survival after progression to CRPC, although multiple options are available for mCRPC. Therefore, there is still a need to improve the therapeutic effect for mCRPC.

Many studies have shown that metabolic syndrome and its components are associated with increased development and progression of aggressive prostate cancer. Metformin, a common well-tolerated oral biguanide prescribed for type II diabetes, could be used to decrease the risk of prostate cancer development and improve the efficacy of treatment. Some studies reported that metformin could enhance the effectiveness of ADT, and improve recurrence-free survival, overall survival and cancer-specific survival. A prospective randomized study reported that metformin potentially lengthen time to CRPC in advanced prostate cancer patients when combined with ADT especially in those with high risk localized prostate cancer, clinically node positive and in those with low tumor volume metastatic hormone-sensitive patients.

After extensive research, there is no published results from prospective randomized trials evaluating the effect of metformin in combination with ADT and abiraterone among patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and newly diagnosed metastatic hormone-sensitive adenocarcinoma of the prostate without small cell carcinoma or small cell components.
* Metastatic adenocarcinoma of the prostate proved by imaging (CT/MRI and/or bone scan).
* Patients must meet the criteria of CRPC.
* No prior treatment with chemotherapy and new-generation hormonal therapy including abiraterone, enzalutamide, apalutamide.
* Patient must give written informed consent before registration and prior to any trial related investigations.
* Age ≥18 years.
* Serum potassium ≥3.5mmol/ L.
* ECOG performance status 0-2
* Ongoing androgen deprivation therapy with drugs or bilateral orchiectomy, and continuous abiraterone plus prednisone.
* Patient agrees not to father a child during participation in the trial and during 3 months thereafter.
* Patient agrees not to participate other interventional trials.
* Patients are able to swallow study drug as whole tablet.

Exclusion Criteria:

* Diagnosed diabetes or fasting blood-glucose ≥ 6.1mmol/L, or glycosylated hemoglobin ≥ 5.6%.
* Previous malignancy within 2 years prior to randomization, with the exception of localized non-melanoma skin cancer and Ta bladder cancer.
* Major surgery within 4 weeks prior to randomization.
* Treatments with 5a-reductase inhibitors, estrogen, cyproterone acetate, and androgen within 4 weeks prior to randomization.
* Known or suspected Central nervous system CNS metastases or active leptomeningeal disease.
* Equivalent dosage of >10mg/day prednisone of glucocorticoids for the treatment of prostate cancer within 4 weeks prior to randomization, or treatment with glucocorticoids for other reasons.
* Prior treatment for prostate cancer with flutamide, bicalutamide, ketoconazole, abiraterone, enzalutamide, apalutamide, docetaxel chemotherapy, or other interventional drugs for prostate cancer.
* Neutrophils < 1.5 x 109/L, platelets < 75 x 109/L, hemoglobin < 100 g/L.
* ALT and AST ≥ 2.5 x ULN, bilirubin ≥ 1.5 x ULN.
* eGFR<45 ml/min/1.73m2.
* Allergic to metformin or any ingredients of this tablet.
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis. Albumin< 30 g/L.
* Clinically significant cardiovascular disease including:
* Myocardial infarction within 6 months prior to randomization.
* Uncontrolled angina within 3 months prior to registration.
* Congestive heart failure NYHA class III or IV.
* History of clinically significant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation, torsades de pointes).
* History of Mobitz II second or third degree heart block without a permanent pacemaker in place.
* Systolic pressure< 86 mmHg.
* Bradycardia, heart rate<45/min.
* Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg OR diastolic blood pressure > 105 mmHg.
* Prior treatment with metformin after diagnosis of prostate cancer.
* Allergic to metformin or any drugs used in this trial.
* Serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. uncontrolled or acute severe infection, uncontrolled diabetes).
* Active or symptomatic viral hepatitis or chronic liver disease. History of pituitary or adrenal dysfunction.
* Gastrointestinal disorder affecting absorption.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-06-23 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival defined from randomization to time till biochemical progression or radiographic progression | start of treatment to disease progression, up to 36 months

SECONDARY OUTCOMES:
Overall survival defined from randomization until death due to any reason | start of treatment to death, up to 36 months
Radiographic progression-free survival defined from randomization until radiographic progression | start of treatment to radiographic progression, up to 36 months
Adverse events which will be assessed according to NCI-CTC AE 5.0 | start of treatment to study completion, up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Yonghong Li, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No